CLINICAL TRIAL: NCT07073573
Title: The Relationship Between Pulpal Biomarker Levels and the Success of Vital Pulp Therapy: A Prospective Clinical Study
Brief Title: Evaluation of Pulpal Biomarkers in Vital Pulp Therapy
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: ertuğrul karataş (Other)
Responsible Party: Sponsor-Investigator, ertuğrul karataş, Associate Professor of Endodontics, Ataturk University
Organization: Ataturk University (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: B.30.2.ATA.0.01.00/535; NO-FUNDING-TRIAL-2025 (Other: University-Sponsored Non-Funded Trial)
Record Dates: First submitted 2025-07-10; First posted 2025-07-18 (Actual); Last update posted 2025-07-20 (Actual); Status verified 2025-07

CONDITIONS: Reversible Pulpitis; Irreversible Pulpitis; Vital Pulp Therapy; Dental Pulp Diseases
Keywords: Pulpal Biomarkers; Vital Pulp Therapy; Inflammatory Cytokines; Dental Pulp Inflammation; Clinical Success; Biomarker Expression
MeSH Terms: conditions — Dental Pulp Diseases | interventions — Pulpotomy

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to one of two parallel arms based on clinical diagnosis: reversible pulpitis or irreversible pulpitis
Who Masked: Participant
Masking Description: Participants were blinded to their group assignment, but investigators were aware of the clinical group classification.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- reversible pulpitis (Active Comparator): Patients diagnosed with reversible pulpitis and treated accordingly
  Interventions: Procedure: Vital pulp therapy
- Irreversible Pulpitis (Active Comparator): Patients diagnosed with irreversible pulpitis and treated accordingly
  Interventions: Procedure: Vital pulp therapy

INTERVENTIONS:
Procedure: Vital pulp therapy — Vital pulp therapy was performed using a calcium silicate-based material after caries removal and coronal pulp exposure. Hemostasis was achieved using sodium hypochlorite before placing the material. Permanent restoration was completed in the same session. Pulpal fluid samples were collected before the intervention to assess biomarker levels. The relationship between biomarker expression and the clinical success or longevity of the treated teeth was evaluated over time
  Other Names: Partial pulpotomy; Pulpotomy

SUMMARY:
This prospective clinical study aims to evaluate the association between the levels of selected pulpal biomarkers and the clinical success of vital pulp therapy in permanent teeth. Patients undergoing vital pulp therapy will be monitored over time, and biomarker expression levels will be analyzed in relation to treatment outcomes. The study intends to provide insight into the predictive value of pulp tissue biomarkers for long-term success in vital pulp procedures.

DETAILED DESCRIPTION:
The aim of this study is to identify the biomarkers that influence the success of vital pulp therapy (VPT), a treatment that offers several advantages over conventional root canal therapy. The study also aims to evaluate the success of VPT in teeth diagnosed with irreversible pulpitis. The success of VPT largely depends on the accurate assessment of pulpal status.

This prospective clinical study will be conducted on 50 patients who apply to the Department of Endodontics, Faculty of Dentistry, Atatürk University, and meet the inclusion criteria. Informed consent will be obtained from all participants. A specially designed clinical assessment form will be completed for each patient to record clinical findings prior to the procedure.

Local anesthesia will be administered using 1.8 mL of 4% articaine with 1:100,000 epinephrine. Following anesthesia, the teeth will be isolated using a rubber dam. Caries removal will be performed under an operating microscope (OPMI) using a diamond bur and aerator. All infected dentin will be removed selectively until hard dentin is reached.

Pulpal bleeding will be controlled by applying a cotton pellet moistened with sterile saline into the cavity for one minute. Subsequently, pulpal fluid and blood samples will be collected using 5 mm-long sterile paper points to ensure equal sample volume per case. Each sample (one per patient) will be transferred into separate sterile Eppendorf tubes containing 500 µL of phosphate-buffered saline (PBS) and stored at -80°C until biochemical analysis. Total bleeding time will be recorded using a chronometer.

The first tube will be used for the analysis of mediators including RANTES (CCL5), MCP-1, TNF-α, TGF-β, IL-1β, TIMP-1, MMP-12, and MMP-1. The second tube will be used to measure MDA, SDA, TAS, and TOS levels.

After sample collection, the exposed pulp will be disinfected with a cotton pellet soaked in 2.5% sodium hypochlorite for 30 seconds. The cavity will then be rinsed with sterile saline and dried. The exposed pulp will be capped with Mineral Trioxide Aggregate (MTA) according to the manufacturer's instructions, and permanent restoration of the tooth will be completed.

Patients will be recalled for follow-up evaluations at 3, 6, and 12 months, during which pulpal vitality will be assessed. A correlation will be established between biomarker levels and clinical success of the vital pulp therapy.

ELIGIBILITY:
Inclusion Criteria:

* Permanent teeth diagnosed with reversible pulpitis
* Patients diagnosed with irreversible pulpitis but without apical radiolucency
* Teeth showing a normal response to cold testing (carbon dioxide snow)
* Teeth with irreversible pulpitis demonstrating prolonged response to cold testing
* Teeth with no sensitivity to percussion or chewing
* In teeth with exposed pulp tissue, bleeding time less than 5 minutes
* In irreversible pulpitis cases, bleeding time less than 10 minutes
* No widening of the periodontal ligament space (periapical index [PAI] ≤ 2)
* Radiographic evidence of deep dentinal caries

Exclusion Criteria:

* Teeth with a negative response to cold testing (carbon dioxide snow)
* Presence of apical radiolucency (PAI > 2)
* Condensed apical periodontitis
* Internal or external root resorption
* History of dental trauma
* Longitudinal root fracture
* Presence of periodontal-endodontic lesions on the day of treatment
* Functional loss (e.g., Grade 3 tooth mobility)
* Swelling associated with the treated tooth
* Teeth that cannot be treated under rubber dam isolation
* Teeth from which less than 2.5 mL of pulpal blood can be collected
* Immunocompromised individuals
* Pregnant women at the time of treatment
* Use of antibiotics, bisphosphonates, or statins within 4 weeks prior to treatment

Ages: 16 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2025-07-25 (Estimated); Study Completion 2026-08-03 (Estimated)

PRIMARY OUTCOMES:
Clinical success of treated teeth with Vital Pulp Therapy | 6-12 months after treatment
  Clinical and radiographic success will be defined as the absence of symptoms (e.g., spontaneous pain, swelling), no sinus tract, no pathological mobility, and no periapical radiolucency. In addition, a positive response to pulp vitality tests (e.g., cold test or EPT) will be considered as an indicator of maintained pulpal vitality.

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk University, Faculty of Dentistry, Department of Endodontics, Erzurum, Erzurum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Iaculli F, Rodriguez-Lozano FJ, Briseno-Marroquin B, Wolf TG, Spagnuolo G, Rengo S. Vital Pulp Therapy of Permanent Teeth with Reversible or Irreversible Pulpitis: An Overview of the Literature. J Clin Med. 2022 Jul 11;11(14):4016. doi: 10.3390/jcm11144016. PMID 35887779
- [Background] Asgary S, Nosrat A. Vital Pulp Therapy: Evidence-Based Techniques and Outcomes. Iran Endod J. 2025;20(1):e2. doi: 10.22037/iej.v20i1.47141. Epub 2025 Jan 1. PMID 39935864